CLINICAL TRIAL: NCT05397054
Title: Community-based Intervention for Monitoring of Salt Intake in Hypertensive Patients
Brief Title: Intervention for Monitoring of Salt Intake in Hypertensive Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: World Health Organization (Other); Thai health promotion foundation. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COA. MURA2021/1004
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Hypertension; Salt; Excess
Keywords: hypertension; salt; salt reduction
MeSH Terms: conditions — Hypertension | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigator (Experimental): Education, Reformulation, Environmental change, Used salt meter
  Interventions: Behavioral: Education; Behavioral: Reformulation; Behavioral: Environmental change; Device: Salt meter
- Control (Active Comparator): standard treatment with standard education
  Interventions: Behavioral: standard treatment

INTERVENTIONS:
Behavioral: Education — - Education: Education about risk of high sodium intake, type of sodium, nutrition ingredients
  Arms: Investigator
Behavioral: Reformulation — - Reformulation: Dietary recommendation in low sodium intake
  Arms: Investigator
Behavioral: Environmental change — - Environmental change: Encourage about low sodium intake in community
  Arms: Investigator
Device: Salt meter — - Used salt meter: at least 3 times/wk
  Arms: Investigator
Behavioral: standard treatment — standard treatment
  Arms: Control

SUMMARY:
Sodium is an essential nutrient for humans, but excessive sodium consumption is causally associated with high blood pressure and increase risk of cardiovascular diseases. Dietary sodium consumption of greater than the recommended daily amount of 5 grams of salt or 2,000 mg of sodium is a major risk factor for CVD-related mortality. From recent national survey, Thai people had consumed more than 9.1 g of salt per day, which was nearly two times above WHO reference level. Dietary salt reduction was unsuccessful because of lacking awareness, and the higher threshold to detect salt taste in chronic high salt ingestion. To create awareness in the community, we should be educated, managed the environmental for salt reduction, and used salt meter to detect sodium content in daily food. This study aimed to compare the efficacy of intervention; education, reformulation, environmental change and used salt meter compared with standard treatment alone in terms of salt intake reduction and blood pressure.

DETAILED DESCRIPTION:
A randomized-controlled trial was conducted in adult 18-70 years old with hypertensive patients (SBP>130 mmHg) in Uthaithani. Participants were randomized to intervention groups (education, reformulation, environmental change and used salt meter) and control group (standard education and treatment). Trial was followed up for 12 weeks. The primary objective was change in 24-hour urinary sodium excretion between groups and secondary objectives was change in systolic and diastolic blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-70 years of age with hypertension
* Systolic blood pressure > 130 mmHg
* Provided informed consent to participate in the study

Exclusion Criteria:

* Participants with end stage kidney disease
* History of adjust antihypertensive agents or diuretic within 2 weeks before enrollment
* Pregnant or breastfeeding women
* Adjustment of any antihypertensive agents during study period
* Participants with salt supplement

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 240 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
24-hour urine sodium excretion | 12 weeks
  Compare the change of 24-hour urine sodium excretion between intervention group, received education, reformulation, environmental change and monitoring of salt intake by salt meter and control group, received standard treatment

SECONDARY OUTCOMES:
blood pressure | 4, 8 12 weeks
  Compare the change systolic and diastolic blood pressure between intervention group, received education, reformulation, environmental change and monitoring of salt intake by salt meter and control group, received standard treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

REFERENCES:
- [Derived] Sonuch P, Aekplakorn W, Pomsanthia N, Boonyagarn N, Makkawan S, Thongchai S, Tosamran W, Kunjang A, Kantachuvesiri S. Community-based intervention for monitoring of salt intake in hypertensive patients: A cluster randomized controlled trial. PLoS One. 2024 Nov 22;19(11):e0311908. doi: 10.1371/journal.pone.0311908. eCollection 2024. PMID 39576798